CLINICAL TRIAL: NCT06808022
Title: Influence of Pre-operative Back Muscle Exercise on Post-operative Outcomes After Spine Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Bahar Shahidi, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 803198
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Spine Pain; Spine Surgery
Keywords: Prehabilitation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/Standard of Care (No Intervention): Standard of Care preoperatively per surgeon recommendation
- Preoperative Resistance exercise (Experimental): Resistance based exercise targeting the back muscles above where the intended surgery is planned
  Interventions: Behavioral: Preoperative Resistance Exercise

INTERVENTIONS:
Behavioral: Preoperative Resistance Exercise — Participants will have been deemed to be medically safe to participate in exercise-based physical therapy based on their physician recommendation and may also undergo an in-person evaluation by a licensed physical therapist to evaluate their physical capacity. This will inform the frequency and intensity of exercise prescription according to a participant's identified physical impairments and activity tolerance levels. Based on this information, an exercise program will be implemented either via web-based HIPAA compliant platforms (e.g. Zoom or WebEx) or in the clinic(e.g if the participant does not have internet access) on a 1-2x/week basis for the 4-6 week pre-operative duration. Each exercise session will be approximately 30 minutes. During these sessions, exercises including gravity-assisted, body-weighted, or body-weight-augmented resistance exercises targeting the paraspinal extensor muscles (multifidus, erector spinae, latissimus dorsi, lower trapezius) will be performed at a mo
  Arms: Preoperative Resistance exercise

SUMMARY:
The purpose of this research study is to gather more information about how improving back muscle function before surgery might influence what happens to the spine and function after surgery. This may assist in developing ways to improve surgical outcomes and determine the benefit of pre-operative exercise, if any.

DETAILED DESCRIPTION:
The investigators intend to enroll patients from UCSD spine clinic. The investigators will include patients who are indicated for a spine surgery. Once participants are identified to be surgical candidates, and have an estimated surgical date that is 4-6 weeks from identification, the participants may undergo pre-operative procedures including a pre-operative evaluation and treatment by a physical therapist, data collection (demographics, medical history, etc.), and filling out relevant questionnaires. Patients will undergo their surgery as scheduled with the spine surgeon as part of their planned standard care unless the surgeon decides that the surgery is no longer necessary. Participation in research does not influence the surgeon's decision. Post-operatively, participants may be asked to undergo a post-operative evaluation and fill out questionnaires.

Upon identification of eligibility, participants may be randomized to one of two study arms using a random number generator. If group characteristics are observed to be unbalanced using this approach, participants may be matched according to demographic or surgical features:

1. Pre-habilitation treatment arm
2. Standard of Care arm Participants in the standard of care arm will undergo all pre-operative activities recommended by their surgeon as per standard care.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals undergoing spinal surgery
* Individuals who have been deemed medically safe to participate in an exercise-based physical therapy program

Exclusion Criteria:

* - Individuals with comorbid conditions or spinal injury inappropriate for participating in an exercise-based physical therapy program as determined by the surgeon (e.g. unstable vertebral fracture)
* Individuals that do not have the ability to commit to the therapy schedule either in-clinic or using the web-based interface
* Non-english speaking individuals (some questionnaires are validated only in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Revision | 1 year
  Patient requires surgical revision within 1 year of index surgery

SECONDARY OUTCOMES:
Length of stay | 3 months
  Postoperative hospital length of stay
Numeric Pain Rating Scale | 1 year
  Numeric Pain Rating Scale for back and leg pain on a 0-10 scale, with 10 being worst pain imaginable and 0 being no pain
Disability | 1 year
  Oswestry Disability Index, in percent, from 0-100. 0 indicating 0% disabled from back pain, and 100% indicating complete disability due to back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided